CLINICAL TRIAL: NCT06736574
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Trial to Assess Efficacy and Safety of Omecamtiv Mecarbil in Patients With Symptomatic Heart Failure With Severely Reduced Ejection Fraction (COMET-HF)
Brief Title: Study With Omecamtiv Mecarbil (CK-1827452) to Treat Chronic Heart Failure With Severely Reduced Ejection Fraction
Acronym: COMET-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 1033; 2024-519219-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: CK-1827452; omecamtiv mecarbil
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omecamtiv Mecarbil (Experimental): Participants randomized to omecamtiv mecarbil will be dosed based on their omecamtiv mecarbil plasma concentration at 25, 37.5 or 50 mg twice daily until at least 850 participants experience a HF event or CV death, whichever comes first.
  Interventions: Drug: Omecamtiv Mecarbil (OM)
- Placebo (Placebo Comparator): Participants randomized to placebo will receive placebo twice daily until at least 850 participants experience a HF event or CV death, whichever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omecamtiv Mecarbil (OM) — Oral Tablet
  Arms: Omecamtiv Mecarbil
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if the investigational drug called omecamtiv mecarbil can reduce the risk of the effects of heart failure, like hospitalization, transplantation, or death in patients with heart failure and severely reduced ejection fraction.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of omecamtiv mecarbil in reducing the risk of the primary composite endpoint of cardiovascular (CV) death, first heart failure (HF) event, left ventricular assist device (LVAD) implantation, cardiac transplantation, and stroke in patients with symptomatic heart failure with severely reduced ejection fraction (HFrEF).

Eligible patients will be randomized 1:1 to investigational product (IP) - omecamtiv mecarbil or placebo. The study is event-driven and will conclude when at least 850 participants experience a HF event or CV death, whichever comes first. An interim analysis for futility and efficacy based on the primary composite endpoint is planned when approximately 570 (67%) of the planned 850 first HF events or CV deaths are observed.

Estimated duration of participation: Up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who meet all the following criteria at screening may be included in the study:

* Are between ≥ 18 years and ≤ 85 years at the signing of informed consent
* Have a history of chronic HFrEF, defined as requiring treatment for HF for a minimum of 3 months prior to screening
* Are receiving oral loop diuretics
* Patients without AFF on screening ECG:

  * LVEF < 30% within 6 months of screening
  * Elevated N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) ≥ 1000 pg/mL (BNP ≥ 300 pg/mL)
* Patients with AFF on screening ECG:

  * LVEF < 25% within 6 months of screening
  * Elevated N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) ≥ 3000 pg/mL (BNP ≥ 900 pg/mL)
  * Not currently taking digoxin
* Are currently hospitalized with the primary reason of HF, or had an HF event within 6 months prior to screening
* Are established on regional standard-of-care HF therapies for at least 30 days prior to screening
* Systolic blood pressure ≤ 130 mmHg and diastolic blood pressure ≤ 90 mmHg

Exclusion Criteria:

Any of the following criteria will exclude potential patients from the study:

* Have AFF on the screening ECG and are currently taking digoxin
* Have had acute coronary syndrome, cardiac surgery, valve surgery, any coronary revascularization, and/or cardiac resynchronization therapy within 3 months of screening
* Are admitted to a long-term care facility or hospice
* Have a projected survival of < 12 months due to non-cardiovascular causes based on clinical judgment
* Are receiving intravenous inotropes or intravenous vasopressors ≤ 3 days prior to screening
* Are receiving mechanical hemodynamic support or mechanical ventilation ≤ 7 days prior to screening
* Are receiving intravenous diuretics, intravenous vasodilators, or supplemental oxygen therapy ≤ 12 hours prior to screening
* Have an estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2 or receiving dialysis at screening
* Have previously had a solid organ transplant
* Are receiving treatment in another investigational device or drug study or are within 30 days of ending such investigational treatment at screening
* Have previously received omecamtiv mecarbil
* Are pregnant or planning pregnancy during the study period, or planning to breastfeed during treatment with IP or within 5 days after the end of treatment with IP

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to the first of event of CV death, HF event, LVAD implantation/cardiac transplantation, or stroke | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Efficacy of omecamtiv mecarbil compared with placebo on the risk of HF outcomes in patients with symptomatic HFrEF and severely reduced ejection fraction in the setting of guideline-directed medical therapy per local standard of care.

SECONDARY OUTCOMES:
Time to the first event of CV death or HF event | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of CV death and HF event
Time to the first HF hospitalization | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of HF hospitalization
Time to the first event of CV death, HF event, LVAD implantation/cardiac transplantation, or stroke in a subgroup of patients with severe HF | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of HF outcomes in patients with severe HF, defined as patients with NYHA class 3-4 symptoms and a HF event within the last 3 months
Time to the first event of CV death, LVAD implantation/cardiac transplantation, or stroke | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of irreversible morbidity/mortality related to HFrEF
Time to CV death | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of CV mortality
Time to first event of stroke | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of stroke
Time to all-cause death | From randomization to the first event of CV death or HF event, whichever occurs first, assessed until the last patient exits the study, estimated to last about 3 years
  Effect of omecamtiv mecarbil compared with placebo on risk of all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Director — Cytokinetics
Locations (181):
- United States (88):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pima Heart and Vascular Clinical Research, Tucson, Arizona
  - National Heart Institute, Beverly Hills, California
  - UC San Diego Health - Sulpizio Cardiovascular Center, La Jolla, California
  - Nutrition Research Center (SPH), Loma Linda, California
  - Keck Medical Center of USC (outpatient clinic), Los Angeles, California
  - UCLA Medical Center Cardiovascular Clinic, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sutter Institute for Medical Research (SIMR), Sacramento, California
  - UC Davis Health, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - California Pacific Medical Center Van Ness Campus, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Stanford University Hospital / Stanford Health Care, Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor - UCLA Medical Center, Torrance, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Cardiology Associates of Fairfield County, P.C, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Health Heart & Vascular Center Outpatient Services, New Haven, Connecticut
  - CHF Heart Clinical (Subject Visits & IP Shipments), Clearwater, Florida
  - Holy Cross Medical Group - Cardiology Associates, Fort Lauderdale, Florida
  - South Florida Research Solutions, LLC, Hollywood, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Broward Research Center, Miami Beach, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - AdventHealth, Orlando, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - The Queen's Medical Center - Punchbowl, Honolulu, Hawaii
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC., Munster, Indiana
  - Deaconess Heart Group, Newburgh, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - AHMG Cardiology and Surgery, Overland Park, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Eastern Main Medical Center dba Northern Light Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Midwest Heart and Vascular Specialists, LLC, Independence, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University Center for Advanced Medicine, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Monmouth Cardiology Associates, LLC, Eatontown, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center / New York - Presbyterian, New York, New York
  - Montefiore Medical Center (Moses Campus), The Bronx, New York
  - WakeMed Heart & Vascular - Cary Cardiology, Cary, North Carolina
  - Clinical and Translational Research Center - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Moses H. Cone Memorial Hospital Operating Corporation d/b/a Cone Health, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - K&R Research LLC, Marion, Ohio
  - University of Hospitals North Ohio Heart, Sandusky, Ohio
  - Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania (University of Pennsylvania School of Medicine), Philadelphia, Pennsylvania
  - Medical University of South Carolina - Gazes Research Institute, Charleston, South Carolina
  - Monument Health Clinical Research, a department of Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Medresearch Inc, El Paso, Texas
  - University of Texas Medical Branch - UTMB, Galveston, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Baylor Scott & White Medical Center- The Hearth Hospital, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Advanced Heart Disease and Transplant, Spokane, Washington
  - Medical College of Wisconsin / Froedtert Hospital, Milwaukee, Wisconsin
- Canada (14):
  - Mazankowski Alberta Heart Institute / University of Alberta Hospital, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - SMH - Cardiology Clinical Trials Inc., Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Oakville Trafalgar Memorial Hospital - Halton Healthcare, Oakville, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
- France (10):
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Haute-Garonne
  - Polyclinique Vauban, Valenciennes, Hauts-de-France
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire Grenoble Alpes - Site Nord Michallon, La Tronche, Isère
  - CHU de Montpellier- Hôpital Arnaud de Villeneuve, Montpellier, Occitanie
  - L'Hôpital Privé Du Confluent, Nantes, Pays de la Loire Region
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer (C.H.I.T.S), Toulon, Var
  - Hôpital Lariboisière - APHP, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
  - APHP - Hôpital Bichât, Paris, Île-de-France Region
- Germany (13):
  - LMU Klinikum - Medizinische Klinik und Poliklinik I, München, Bavaria
  - Universitätsklinik Würzburg Deutsches Zentrum für Herzinsuffizienz, Würzburg, Bavaria
  - Helios Klinikum Erfurt GmbH, Erfurt, Germany
  - Universitaetsklinikum Jena, Jena, Germany
  - Marienhaus Klinikum Mainz GmbH, Mainz, Germany
  - UKE, Klinik fur Kardiologie, Hamburg, Hamburg
  - UKE, Klinik für Kardiologie, Hamburg, Hamburg
  - Kerckhoff-Klinik GmbH, Bad Nauheim, Hesse
  - Universitaetsklinikum Frankfurt, Med. Klinik III - Kardiologie, Angiologie, Frankfurt am Main, Hesse
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen, Hesse
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Dr. med. Jens Taggeselle, Markkleeberg, Saxony
- Greece (9):
  - General Hospital of Athens ''G. Gennimatas'', Athens, Attica
  - General Hospital of Athens ''Hippokratio'', Athens, Attica
  - General Hospital of Nea Ionia ''Konstantopouleio-Patision'', Athens, Attica
  - University General Hospital ''ATTIKON'' - General Hospital of West Attica H, Chaïdári, Attica
  - General Hospital ''Asklepieio Voulas'', Voula, Attica
  - University General Hospital of Alexandroupolis, Alexandroupoli, Evros
  - University General Hospital of Larissa, Larissa, Larissa
  - Papageorgiou General Hospital of Thessaloniki, Efkarpia, Thessaloniki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki, Thessaloniki
- Italy (9):
  - ASST Spedali Civili di Brescia, Brescia, BS
  - Ospedale Infermi, Rimini, Emilia-Romagna
  - Ospedale di Arzignano, Arzignano, Lombardy
  - Centro Cardiologico Monzino, Milan, Lombardy
  - IRCCS Multimedica, Sesto San Giovanni, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, MI
  - A.O. Perugia - Ospedale S.Maria della Misericordia, Perugia, Province of Perugia
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant' Anna, Cona
  - IRCCS San Raffaele, Roma
- Poland (12):
  - Balsammedica Sp. z o.o., Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny UCK WUM, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Krakowski Szpital Specjalistyczny im. Sw. Jana Pawla II, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 2 UM w Lodzi, Lodz
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Szpital Sw. Anny w Miechowie, Miechów
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Poradnia AKA-MED Centrum Sp. z o.o., Ruda Śląska
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - Wojewodzki Szpital Zespolony im. L. Rydygiera, Torun
- Spain (17):
  - Hospital Universitario A Coruña, A Coruña, A Coruña
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital San Juan de la Cruz, Úbeda, Jaen
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Valencia
- United Kingdom (9):
  - Harefield Hospital, Harefield, Greater London
  - Southampton General Hospital, Southampton, Hampshire
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Castle Hill Hospital, Cottingham
  - Russells Hall Hospital, Dudley
  - Ulster Hospital, Dundonald
  - Glasgow Royal Infirmary, Glasgow
  - Great Western Hospitals, Swindon

IPD SHARING:
Plan to Share IPD: No